CLINICAL TRIAL: NCT00000268
Title: Cocaine Abuse and Attention Deficit Disorder
Brief Title: Cocaine Abuse and Attention Deficit Disorder - 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: New York State Psychiatric Institute (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: NIDA-09236-3; P50-09236-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion

SUMMARY:
The purpose of this study is to evaluate cocaine abuse and Attention Deficit Disorder

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of methylphenidate and bupropion in treating individuals with adult Attention Deficit Disorder.

ELIGIBILITY:
Inclusion Criteria:

current adult ADHD current cocaine dependence

Exclusion Criteria:

no current major depression

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 1995-05; Study Completion 1998-11

PRIMARY OUTCOMES:
Side effects
Craving
Drug use
ADHD symptoms
Improvement in functioning
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States